CLINICAL TRIAL: NCT05961826
Title: National Cohort About Epidemiology, Clinical and Genetic Heterogeneity of the "Low-Phospholipid-Associated Cholelithiasis" (LPAC) Syndrome
Brief Title: COLPAC (RaDiCo Cohort) (RaDiCo-COLPAC)
Acronym: COLPAC
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-14
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Low Phospholipid Associated Cholelithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to describe the various clinical, biological and radiological manifestations of LPAC syndrome, defined according to standard diagnostic criteria, or according to criteria extended to all symptomatic recurrent biliary lithiasis, and delineate the various possible evolutions.

Participants will be followed for 5 years and the inclusion sites will collect the necessary data at least once a year as part of routine patient care. A quality of life self-questionnaire will be completed by participants during these visits.

ELIGIBILITY:
Inclusion Criteria:

* Children or adults meeting the standard* or extended** diagnostic criteria for LPAC syndrome:

  1. First symptoms before the age of 40 years
  2. Radiological images compatible with the existence of intrahepatic lithiasis
  3. Recurrence of symptoms after cholecystectomy

     (*) standard criteria: symptomatic biliary lithiasis with at least 2 out of 3 criteria

     (**) extended criteria: symptomatic biliary lithiasis with 1 out of 3 criteria

     Exclusion Criteria:
* Patients who have undergone liver transplantation

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study concerns all prevalent and incident patients who meet the standard or extended diagnostic criteria for LPAC syndrome, whatever the existing genetic data concerning ABCB4, or who have been referred as having a mutation in the ABCB4 gene in a clinical context of biliary lithiasis.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of the clinical manifestations of LPAC syndrome like personal and family medical history of the disease, clinical features, medical complications, co-morbidities, death (age of onset and cause). | Through study completion, an average of 5 years
Descriptive analysis of the biological manifestations of LPAC syndrome like hepatic biochemical tests and glucido-lipid tests | Through study completion, an average of 5 years
Descriptive analysis of the radiological manifestations of LPAC syndrome like presence of stones or signs of intrahepatic, vesicular or main bile duct micro-lithiasis | Through study completion, an average of 5 years

SECONDARY OUTCOMES:
Description of diagnostic practices by a descriptive analysis of sequences of medical procedures used to diagnose LPAC syndrome. | Through study completion, an average of 5 years
Description of therapeutic practices by a descriptive analysis of the different curative and symptomatic treatments offered depending on the stage of the disease and the type of extra-hepatic complications. | Through study completion, an average of 5 years
Description of patient management practices. | Through study completion, an average of 5 years
Identification of new diagnostics by refining the collection of semiological fields of 1st degree relatives and including patients with recurrent symptomatic biliary lithiasis who do not fully meet the current diagnostic criteria for LPAC syndrome | Through study completion, an average of 5 years
  The extension of the criteria will be proposed on the basis of the collection of all the semiological fields of patients diagnosed with an LPAC syndrome defined according to the usual or extended criteria and their 1st degree relatives.
  The extended diagnostic criteria are :
  * Age of onset of the disease over 40 years of age
  * The presence of recurrent biliary lithiasis without radiological signs characteristic of LPAC syndrome (comet tails or intrahepatic lithiasis).
  Patients with symptomatic gallstones who have only one of the 3 criteria for LPAC syndrome (onset before the age of 40, intrahepatic microlithiasis, recurrence after cholecystectomy).
Evaluation of response to medical and interventional treatments. | Through study completion, an average of 5 years
  This evaluation criterion will be the search for correlation between response or non-response to medical and interventional treatments. This will be analysed by looking at the presence or absence of certain clinical, biochemical, molecular and radiological features of the disease such as :
  * No reduction in the frequency or intensity of painful attacks.
  * No reduction in the number of complications.
  * No improvement or normalisation of liver tests.
  * No regression or disappearance of radiological signs of intrahepatic lithiasis
  * No improvement in the criteria for assessing quality of life and impact on social life
Identification of prognostic factors (clinical, biochemical, radiological) associated with a poor therapeutic response by assessing the occurrence of events such as : - Fatal or non-fatal complications - Death due to hepatic or other causes | Through study completion, an average of 5 years
Assessing the impact of LPAC syndrome on quality of life. | Through study completion, an average of 5 years
  Impact of disease on quality of life will be evaluated through scores of quality of life questionnaires (SF-36)
Evaluation of the proportion of patients referred to LPAC within the population referred to the hepatology and/or digestive surgery departments for biliary lithiasis during the same study period | Through study completion, an average of 5 years
  The relative prevalence of LPAC syndrome (number of cases of LPAC syndrome compared with the number of cases of gallbladder disease) will be measured from 1 March 2016 to 28 February 2017, based on cases recorded in the centres participating in the study.
  The relative incidence (number of new cases of LPAC syndrome compared with the number of new cases of gallstones) will be measured over the same period, in the same centres.
  The total number of patients seen in hospital or in consultation during the same period for gallstones will be collected in each participating hospital using the pmsi code.

OTHER OUTCOMES:
Deepening the study of the genotype/phenotype correlations of the ABCB4 gene with assessment of the number of painful attacks and complications, presence of radiological signs, measurement of biological assays, good or poor response to treatment | Through study completion, an average of 5 years
Documenting the genetic transmission profile and heritability (penetrance) of the LPAC syndrome by analysing the phenotypes and genotypes of patients and their 1st degree relatives (whether or not they have declared illness). | Through study completion, an average of 5 years
  The evaluation criteria will be :
  * the collection of common genetic mutations in the patient and 1st degree relatives (carried out as part of the diagnostic study of the index case)
  * the search for common phenotypes in the patient and 1st degree relatives (carried out as part of the diagnostic study of the index case)
Search for new susceptibility genes in patients without gene alterations of ABCB4 | Through study completion, an average of 5 years
Search for modulating genes in mutated and non-mutated ABCB4 patients. | Through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CORPECHOT, Principal Investigator — INSERM UMR_S938
Locations (21):
- France (21):
  - Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence
  - Centre Hospitalier Annecy Genevois, Annecy
  - Hôpital Avicenne, Bobigny
  - Hôpital Haut-Lévêque, Bordeaux
  - Hôpital Saint Camille, Bry-sur-Marne
  - Hôpital Côte de Nacre, Caen
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital François Mitterrand, Dijon
  - Hôpital Michallon, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - Centre hospitalier régional d'Orléans, Orléans
  - Hôpital Saint-Antoine, Paris
  - Hôpital Jean Bernard, Poitiers
  - Hôpital Robert Debré, Reims
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Civil, Strasbourg
  - Hôpital Rangueil, Toulouse
  - Hôpital Paul Brousse, Villejuif